CLINICAL TRIAL: NCT04101279
Title: Evaluation of the Effectiveness and Safety of the Midurethral Synthetic Tape With Tension Control Mechanism and Midurethral Tension Free Tape
Brief Title: Midurethral Synthetic Tape With Tension Control Mechanism Versus Midurethral Free Tape
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Gevorg Kasyan, Professor, Moscow State University of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MoscowSUMD
Record Dates: First submitted 2019-06-14; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Urinary Stress Incontinence
Keywords: stress urinary incontinence; midurethral tension free tape; patient reported outcome; bladder outlet obstruction; complications; tension control mechanism
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Bladder Neck Obstruction

STUDY DESIGN:
Intervention Model Description: Randomized controlled comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midurethral synthetic tape with tension control mechanism (Experimental)
  Interventions: Procedure: surgical management of stress urinary incontinence with synthetic tape with tension control mechanism.
- midurethral tension free tape (Active Comparator)
  Interventions: Procedure: surgical management of stress urinary incontinence with midurethral tension free tape.

INTERVENTIONS:
Procedure: surgical management of stress urinary incontinence with midurethral tension free tape. — Standard protocol for the surgical treatment of stress urinary incontinence using a transobturator approach.
  Arms: midurethral tension free tape
Procedure: surgical management of stress urinary incontinence with synthetic tape with tension control mechanism. — Standard protocol for the surgical treatment of stress urinary incontinence using a transobturator approach. A absorbing gasket attached to the middle of the tape provides tension control.
  Arms: Midurethral synthetic tape with tension control mechanism

SUMMARY:
This is a prospective, comparative randomized controled trial. The general purposes of this study is to compare the efficacy and safety of midurethral synthetic tape with tension control mechanism and conventional midurethral tension free tape as surgical treatment for female urinary stress incontinence.

ELIGIBILITY:
Inclusion Criteria:

Women suffering from stress urinary incontinence, mixed urinary incontinence with prevalence stress urinary incontinence

Exclusion Criteria:

* Pregnancy
* Women with neurogenic bladder dysfunction
* Recurrent stress urinary incontinence
* Woman with history of pelvic surgery
* Mixed urinary incontinence with prevalence urgency urinary incontinence
* Women who suffer from advanced POP (POP-Quantification system (POP-Q) stage more than 2)
* Women with acute urinary tract infection
* Women with bladder outlet obstruction
* Women who are not able to give informed consent or participate with this randomized research study for any other reason

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcome measured as urogenital distress inventory (UDI-6) will be assessed before and after surgery at 12 weeks and 1 year. | 1 year
  The UDI measures the impact of urinary incontinence on activities, roles, and emotional states in women. This questionnaire presented six questions related to urinary disorders. The patient could answer "Not at all", "A little bit", "Moderately" or "Greatly", to each of the questions, each answer is evaluated at 0, 1, 2 or 3 points, respectively, and then summed up. The final score means that the greater the sum of the indicators, the worse the patient's condition.
  This score reflects the condition of the patient before and after surgery at 12 weeks and 1 year.

SECONDARY OUTCOMES:
Bladder outlet obstruction measured during urodynamics pressure flow study | 1 year
  When the urodynamic research indicators deviate (Qmax < 12 ml/s and Postvoid residual volume (PVR) > 100 ml, we establish a diagnosis bladder outlet obstruction.
Stress cough test measured before and after surgery. | 1 year
  Objective cure rate will be not the leakage at physical examination cough test with full bladder (200-400ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow state university of medicine and dentistry named after A.I. Evdokimov, Moscow, Russia